CLINICAL TRIAL: NCT01370551
Title: A Clinical Study of Pharmacokinetics, Efficacy and Safety of Vaginal Application of Lyophilised Lactobacilli and 0.03 mg Estriol (Gynoflor®) on Atrophic Vaginitis in Postmenopausal Breast Cancer Patients Treated With Aromatase Inhibitors
Brief Title: Clinical Study of Vaginal Lactobacilli and Estriol (Gynoflor®) for Atrophic Vaginitis in Breast Cancer Patients
Acronym: Gynoflor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medinova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 806109
Record Dates: First submitted 2011-05-10; First posted 2011-06-10 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Atrophic Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Estriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gynoflor (Experimental): Gynoflor vaginal tablets 1/day x 4 weeks, then 3/week for 8 weeks
  Interventions: Drug: Estriol 0.03 mg, lyophylized lactobacillus

INTERVENTIONS:
Drug: Estriol 0.03 mg, lyophylized lactobacillus — Vaginal tablet with lyophilised lactobacilli and 0.03 mg estriol; Once daily for 28 days then 3 times per week for 8 weeks;
  Other Names: Gynoflor

SUMMARY:
The purpose of this study is to assess the long term safety and efficacy of the vaginal application of Gynoflor®, an extremely low dosed estrogen therapy with lactobacilli, on atrophic vaginitis in postmenopausal breast cancer patients who have been treated with aromatase inhibitors.

DETAILED DESCRIPTION:
Two center phase I pharmacokinetic study assessed circulating estrogens in breast cancer patients on a non-steroidal aromatase inhibitor (NSAI) with vaginal atrophy using vaginal ultra-low-dose 0.03 mg estriol (E3) and Lactobacillus combination vaginal tablets (Gynoflor). 16 women on nonsteroidal aromatase inhibitor with severe vaginal atrophy applied a daily vaginal tablet of Gynoflor for 28 days followed by a maintenance therapy of 3 tablets weekly for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with breast cancer on non-steroidal AI therapy (AI therapy start at least 6 months ago, and are scheduled to receive them during the study)
2. Postmenopausal and age ≥52 with cessation of menses for at least 12 months
3. Age 52 - 75 years
4. Clinical symptoms of vaginal atrophy
5. Vaginal pH > 5.0
6. Karnofsky score ≥80%
7. Signed Informed Consent Form together with contractual capability

Exclusion Criteria:

1. Local or systemic use of any other sexual hormones (estrogens, progestins, androgens), 6 months before and during study
2. Local or systemic use of phytoestrogens or products known for or taken to improve vaginal mucosal function, risk of vaginal infections, or vulvovaginal symptoms, 4 weeks before and during study
3. Local or systemic use of any other anti-infectives, 2 weeks before and during study
4. Use of any other vaginal medication, vaginal rinses and/or moisturizers, gels containing xylocain or other analgesic products to decrease pain during intercourse, 1 week before and during study
5. Known or suspected hypersensitivity or intolerance to the study medications, inclusive their excipients
6. Suspicion of or clinically manifest sexually transmitted infections (infections with Neisseria gonorrhoea, Chlamydia trachomatis, Treponema pallidum, genital herpes, Trichomonas vaginalis, genital condylomata, HIV)
7. Clinical evidence of vaginal infections requiring extra treatment
8. Any infections of the upper genital tract
9. Hysterectomy
10. Genital haemorrhage of unknown origin
11. Malignant or pre-cancerous conditions of the uterus, vulva and/or vagina (PAP smear less than 3 years ago)
12. Acute thrombophlebitis, thromboembolic disorders or a history of these disorders in association with previous use of oestrogen preparations
13. Abuse of alcohol or drugs
14. All chronic illnesses which could influence the absorption, distribution, biotransformation or elimination of the test preparation
15. Patient has a condition or is in a situation which, in the investigator's opinion, may put the patient in significant risk, may confound the study result, or may interfere significantly with the patient's participation in the study
16. BMI lower than 18.5 or higher than 30
17. Patient on steroidal AIs (aromasin)
18. Vulvo-dermatological conditions (like Lichen sclerosus, Lichen rubrus, Psoriasis)
19. Genital prolapses
20. Endometriosis
21. Use of antibiotics or chemotherapeuticals which are harmful to lactobacilli
22. Participation of patient in another investigational drug study, with the exception of treatment optimisation studies with non-steroidal aromatase inhibitors (AI)s
23. Previous participation in this study
24. Patient is a relative of, or staff directly reporting to the investigator
25. Patient is an employee of the sponsor

Ages: 52 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Neven, Prof. Dr., Principal Investigator — University Hospital Leuven, Belgium; Stefan Buchholz, PD Dr., Principal Investigator — Department of Obstetrics and Gynaecology, University of Regensburg, Germany; Gilbert Donders, Prof. Dr., Principal Investigator — Femicare, University Hospital, Leuven, Belgium
Locations (2):
- University Hospital Leuven, Leuven, Belgium
- Department of Obstetrics and Gynaecology, University of Regensburg, Regensburg, Germany

REFERENCES:
- [Result] Donders G, Neven P, Moegele M, Lintermans A, Bellen G, Prasauskas V, Grob P, Ortmann O, Buchholz S. Ultra-low-dose estriol and Lactobacillus acidophilus vaginal tablets (Gynoflor((R))) for vaginal atrophy in postmenopausal breast cancer patients on aromatase inhibitors: pharmacokinetic, safety, and efficacy phase I clinical study. Breast Cancer Res Treat. 2014 Jun;145(2):371-9. doi: 10.1007/s10549-014-2930-x. Epub 2014 Apr 10. PMID 24718774
- [Result] Buchholz S, Mogele M, Lintermans A, Bellen G, Prasauskas V, Ortmann O, Grob P, Neven P, Donders G. Vaginal estriol-lactobacilli combination and quality of life in endocrine-treated breast cancer. Climacteric. 2015 Apr;18(2):252-9. doi: 10.3109/13697137.2014.991301. Epub 2015 Jan 20. PMID 25427450
- [Result] Donders G, Bellen G, Neven P, Grob P, Prasauskas V, Buchholz S, Ortmann O. Effect of ultra-low-dose estriol and lactobacilli vaginal tablets (Gynoflor(R)) on inflammatory and infectious markers of the vaginal ecosystem in postmenopausal women with breast cancer on aromatase inhibitors. Eur J Clin Microbiol Infect Dis. 2015 Oct;34(10):2023-8. doi: 10.1007/s10096-015-2447-1. Epub 2015 Jul 30. PMID 26223323
- See also: Publication of main results — https://pubmed.ncbi.nlm.nih.gov/24718774/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gynoflor: Gynoflor vaginal tablet with lyophilised lactobacilli and 0.03 mg estriol:1 x 28 days, then 3x per week x 8 weeks
Period: Overall Study
Arm/Group | Gynoflor
Started | 16 (Enrolled)
Completed | 16 (Analyzed)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Gynoflor: Gynoflor vaginal tablet with lyophilised lactobacilli and 0.03 mg estriol: 1 x 28 days, then 3x per week x 8 weeks
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 57 [52 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 8
  Germany | 8
Estriol [Mean (Standard Deviation); unit: pg/ml] | 104.5 (40.9)
Follicule Stimulating Hormone (FSH) [Mean (Standard Deviation); unit: mIU/ml] | 107.88 (48.62)
Luteinizing hormone (LH) [Mean (Standard Deviation); unit: mIU/ml] | 36.46 (11.05)
Sex hormone binding globulin (SHBG) [Mean (Standard Deviation); unit: nmol/l] | 73.04 (29.66)
Vaginal maturation index (VMI) [Mean (Standard Deviation); unit: %] — The vaginal maturation index (VMI) was based on the percentages of superficial (X3) and intermediate (X2) epithelial cells present in the vaginal smear, and was calculated according to the following formula: VMI= 0.5(X2) + 1(X3)
  % | 31.2 (19.4)
Lactobacillary grade (LBG) [Mean (Standard Deviation); unit: units on a scale] — LBG I Normal Predominantly lactobacillary morphotypes with few coccoid bacteria, LBG IIa Slightly disturbed Slightly disturbed, fairly normal, LBG IIb Moderately disturbed Moderately disturbed, rather abnormal, LBG III Abnormal Abundant other bacteria but no or few Lactobacilli present
  For the analysis, each of the categories were assigned a numeric score (LBG I= 1, LBG IIa= 2, LBG IIb= 3, LBG III= 4) where lower values indicate a better outcome
  units on a scale | 3.9 (0.3)
Bacterial vaginosis (BV) score [Mean (Standard Deviation); unit: units on a scale] — * Score 0: no BV flora present
  * Score 1: partial BV
  * Score 2: full BV
  units on a scale | 0.1 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentrations of Estriol (E3)
Description: Estrogens were analyzed using a highly sensitive gas chromatography-mass spectrometry (GC/MS) method. The lower limits of quantitation (LLOQ) were 10.00 pg/ml for E3, 1.The coefficient of variation (CV, intra-assay variation) was 2.0 % for E3 (calibration range (CR) 10.00-500.00 pg/).
  The lower limits of quantitation (LLOQ) were 1.00 pg/ml for E2, and 2.00 pg/ml for E1.The coefficient of variation (CV, intra-assay variation) was 4.2 % for E2 (CR 1.00-150.00 pg/ml), and 3.4 % for E1 (CR 2.00-300.00 pg/ml).
Time Frame: -0.5, 0.5, 1, 2, 3, 4, 6, 8, 24 hours on days 0 and 28
Measure: Mean (Full Range); unit: pg/ml
Groups:
- Gynoflor: Gynoflor: Vaginal tablet with lyophilised lactobacilli and 0.03 mg estriol; once daily for 28 days then 3 times per week for 8 weeks;
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
pg/ml
  -0.5 h (Day 0) | 0 [0 to 0]
  -0.5 h (Day 28) | 0.91 [0 to 14.5]
  0.5 h (Day 0) | 3.83 [0 to 14.10]
  0.5 h (Day 28) | 1.58 [0 to 12.90]
  1 h (Day 0) | 11.04 [0 to 18.8]
  1 h (Day 28) | 1.55 [0 to 14.40]
  2 h (Day 0) | 72.73 [0 to 168]
  2 h (Day 28) | 1.96 [0.00 to 16.60]
  3 h (Day 0) | 84.35 [0.00 to 160.00]
  3 h (Day 28) | 2.48 [0.00 to 29.20]
  4 h (Day 0) | 28.29 [0.00 to 67.50]
  4 h (Day 28) | 3.12 [0.00 to 37.70]
  6 h (Day 0) | 0.00 [0.00 to 0.00]
  6 h (Day 28) | 7.33 [0.00 to 39.50]
  8 h (Day 0) | 0.00 [0.00 to 0.00]
  8 h (Day 28) | 10.23 [0.00 to 43.70]
  24 h (Day 0) | 0.00 [0.00 to 0.00]
  24 h (Day 28) | 0.00 [0.00 to 0.00]

2. Primary Outcome: Calculation of Pharmacokinetic Parameters Estriol: Cmax
Description: Cmax is the highest measured concentration
Time Frame: Days 0 and 28
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
pg/ml
  Cmax (Day 0) | 104.5 (40.9)
  Cmax (Day 28) | 15.8 (13.9)

3. Secondary Outcome: Baseline / Trough Serum Concentrations of Estriol
Time Frame: Days 0, 14, 28, 56 and 84
Population: PP
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Gynoflor: This study consists only of this arm.
  Gynoflor: Vaginal tablet with lyophilised lactobacilli and 0.03 mg estriol; Once daily for 28 days then 3 times per week for 8 weeks;
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
pg/ml
  Estriol (Day 0) | 0.00 (0.00)
  Estriol (Day 14) | 5.11 (14.01)
  Estriol (Day 28) | 0.91 (3.63)
  Estriol (Day 56) | 0.00 (0.00)
  Estriol (Day 84) | 0.00 (0.00)

4. Secondary Outcome: Vaginal pH
Description: The normal vaginal pH is 3.8-5.0 pH is a logarithmic scale used to specify the acidity or basicity of aqueous solutions. The scale has values ranging from zero (the most acidic) to 14 (the most basic). Pure water has a pH value of 7. This value is considered neutral-neither acidic or basic.
Time Frame: at all visits during 12 weeks
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
pH
  Entry (Day 0) | 6.0 (0.3)
  C1 (Day 14) | 4.6 (0.5)
  C2 (Day 28) | 4.4 (0.4)
  C3 (Day 56) | 4.6 (0.5)
  C4 (Day 84) | 4.5 (0.5)

5. Primary Outcome: Calculation of Pharmacokinetic Parameters Estriol: Tmax
Description: Tmax is the peak time at which the Cmax (maximum concentration) was measured
Time Frame: Days 0 and 28
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
hours
  Tmax (Day 0) | 2.5 (0.5)
  Tmax (Day 28) | 7.2 (1.5)

6. Primary Outcome: Calculation of Pharmacokinetic Parameters Estriol: Area Under the Curve (AUC)
Description: Area under the curve from administration to the last measured concentration (AUC0-24)
Time Frame: Days 0 and 28
Population: PP
Measure: Mean (Standard Deviation); unit: hours * pg/ml
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
hours * pg/ml
  AUC (0-24h) (Day 0) | 212 (93.2)
  AUC (0-24h) (Day 28) | 130.7 (147.2)

7. Secondary Outcome: Baseline / Trough Serum Concentrations of Luteinizing Hormone (LH)
Time Frame: Days 0, 14, 28, 56 and 84
Population: PP
Measure: Mean (Standard Deviation); unit: mIU/ml
Groups:
- Gynoflor: Gynoflor: Vaginal tablet with lyophilised lactobacilli and 0.03 mg estriol; once daily for 28 days then 3 times per week for 8 weeks
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
mIU/ml
  LH (Day 0) | 36.46 (11.05)
  LH (Day 14) | 34.52 (12.18)
  LH (Day 28) | 34.02 (12.68)
  LH (Day 56) | 34.2 (49.87)
  LH (Day 84) | 35.13 (10.34)

8. Secondary Outcome: Baseline / Trough Serum Concentrations of Sex Hormone Binding Globulin (SHBG)
Time Frame: Days 0, 14, 28, 56 and 84
Population: PP
Measure: Mean (Standard Deviation); unit: nmol/ml
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
nmol/ml
  SHBG (Day 0) | 73.04 (29.66)
  SHBG (Day 14) | 74.24 (35.35)
  SHBG (Day 28) | 71.29 (31.88)
  SHBG (Day 56) | 73.35 (32.76)
  SHBG (Day 84) | 72.43 (34.57)

9. Secondary Outcome: Baseline / Trough Serum Concentrations of Follicule Stimulating Hormone (FSH)
Time Frame: Days 0, 14, 28, 56 and 84
Population: PP
Measure: Mean (Standard Deviation); unit: mIU/ml
Arm/Group | Gynoflor
Number analyzed (Participants) | 16
mIU/ml
  FSH (Day 0) | 107.88 (48.62)
  FSH (Day 14) | 103.71 (39.76)
  FSH (Day 28) | 98.94 (34.95)
  FSH (Day 56) | 103.55 (37.53)
  FSH (Day 84) | 105.93 (43.69)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Gynoflor
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 14/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gynoflor (N=16)
Vaginal discharge (Reproductive system and breast disorders) | 5 (7)
cystitis (Renal and urinary disorders) | 3 (3)
Gastro-intestinal disorders (Gastrointestinal disorders) | 3 (5)
Influenza-like ilness (General disorders) | 2 (2)
Ear and Labyrinth disorders (Ear and labyrinth disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The weaknesses of the study were small numbers for testing of some parameters (especially dyspareunia).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes